CLINICAL TRIAL: NCT03146988
Title: Randomised, Double-Blind, Single, 6 mg Fixed Dose, Two Treatment, Two-Period, Two-Sequence, Two-Way Crossover Comparative Pharmacokinetic and Pharmacodynamic (Phase I) Study of RGB-02 Compared to Neulasta® in Healthy Adult Subjects
Brief Title: Study to Compare the Pharmacokinetics and Pharmacodynamics of 6 mg RGB-02 to 6 mg Neulasta
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gedeon Richter Plc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RGB-02-001
Record Dates: First submitted 2017-04-26; First posted 2017-05-10 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Bioequivalence
MeSH Terms: interventions — pegfilgrastim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RGB-02 6 mg SC (test product) (Experimental)
  Interventions: Drug: RGB-02 or Neulasta® (pegfilgrastim)
- Neulasta® (Active Comparator)
  Interventions: Drug: RGB-02 or Neulasta® (pegfilgrastim)

INTERVENTIONS:
Drug: RGB-02 or Neulasta® (pegfilgrastim) — Pre-filled syringe containing 6 mg RGB-02 or Neulasta® in 0.6 mL, administered as subcutaneous injection into the abdominal area

SUMMARY:
Single-centre, double-blind, randomised, two-period, two-way crossover study to investigate the pharmacokinetics and pharmacodynamics of RGB-02 as compared to Neulasta® administered as a single subcutaneous injection in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or non-pregnant, non-lactating healthy females aged 18 to 55 years
* Body mass index ≥19.0 to ≤30.0 kg/m2
* Body weight >55 kg"

Exclusion Criteria:

* Prior exposure to filgrastim, pegfilgrastim or lenograstim (Period 1 only)
* Subjects who have received any IMP in a clinical research study within the previous 3 months
* History of any drug or alcohol abuse in the past 2 years
* Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine)
* Current smokers who smoke more than 10 cigarettes per day
* Positive drugs of abuse test result
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2017-09-14 (Actual); Study Completion 2017-10-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter: AUC0-inf | 67 days
  Area under the serum concentration vs time curve from dosing to the last measured time point
Pharmacokinetic parameter: Cmax | 67 days
Pharmacodynamic parameter: ANCmax | 67 days
Pharmacodynamic parameter: ANC AOBEC0-tlast | 67 days

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Clinical, Ruddington, Nottingham, United Kingdom